CLINICAL TRIAL: NCT03863509
Title: E-Cigarette Effects on Markers of Cardiovascular and Pulmonary Disease Risk (Aka CLUES - Cardiac and Lung E-cig Smoking Study)
Brief Title: E-Cigarette Effects on Markers of Cardiovascular and Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2017-1090; 1R01HL139331-01 (NIH); Protocol Version 4/26/2021 (Other: UW Madison); A534225 (Other: UW Madison); SMPH\MEDICINE\CARDIOLOGY (Other: UW Madison)
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Tobacco Use; E-Cigarette Use; Cardiovascular Diseases; Pulmonary Disease
Keywords: vape; E-Cigarette; E-cig
MeSH Terms: conditions — Tobacco Use; Vaping; Cardiovascular Diseases; Lung Diseases | interventions — Tobacco Products; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Exclusive Smokers: Smokes Daily; >/= 5 cigarettes/day for last 6 months
  Interventions: Behavioral: Cigarettes
- Exclusive E-Cig users: E-cig usage >/= 5 days/week for last 3 months
  Interventions: Behavioral: E-Cigarettes
- Never users: < 100 cigarettes in lifetime, none for > 5 years; < 3 E-cig usage in lifetime

INTERVENTIONS:
Behavioral: Cigarettes — smokes daily
  Groups: Exclusive Smokers
Behavioral: E-Cigarettes — E-cigarette usage >/= 5 days/week
  Other Names: E-cig; Vape
  Groups: Exclusive E-Cig users

SUMMARY:
This study is designed to enhance the understanding of the possible health effects of e-cigarette use by relating the acute and long-term use of e-cigarettes and conventional cigarettes ("products") to well-validated cardiovascular and pulmonary disease biomarkers. Participants will be enrolled in 3 groups: exclusive e-cigarette users, exclusive cigarette smokers, and a control group of never-users. Participants can expect up to 4 weeks of study participation.

DETAILED DESCRIPTION:
E-cigarette use is increasing rapidly in the United States, especially amongst youth, underscoring the vital need to improve understanding of its health risks. Relevant data could inform policy, guide public health and clinical intervention efforts, and inform individuals who might use or who are using this product. This research will significantly enhance the understanding of the possible health effects of e-cigarette use by relating the acute and long-term use of e-cigarettes and conventional cigarettes ("products") to well-validated cardiovascular and pulmonary disease biomarkers. 3 different "use-groups" of participants will be enrolled: exclusive e-cigarette users (n=165), exclusive cigarette smokers (n=165), and a "control" group of never-users (n=110). These groups reflect the primary decisions that people can make regarding their future tobacco use: to continue to smoke cigarettes, to switch to e-cigarettes, or to avoid tobacco use entirely. It is essential that smokers and health care providers have accurate information on the health effect of these choices.

[Additionally, 100 participants will be invited to be part of an epigenetics sub-study (50 E-cig users, 25 smokers and 25 controls), prior to smoking, an additional 16 ml of blood will be collected in Vacutainer cell separation tubes for peripheral blood monocyte (PBMC) Isolation containing sodium citrate.]

Product use will be related to well-validated biomarkers that sensitively and reproducibly reflect mechanisms, injury, and/or future risk related to cardiovascular or pulmonary disease. Biomarkers will be related to: 1) acute product use in the laboratory (exposure challenges), 2) lifetime history of product use, and/or 3) real-time measures of product use in participants' daily lives. The primary cardiovascular biomarkers are brachial artery flow-mediated dilation (a measure of endothelial function) and carotid intima-media thickness, a measure of subclinical arterial injury and atherosclerosis. The primary pulmonary disease biomarkers will be measures of lung volumes and flow rates (Forced Expiatory Volume exhaled in the first second (FEV1), Forced vital capacity (FVC), FEV1/FVC) obtained by spirometry. Treadmill exercise stress testing will be performed (to assess aerobic fitness), electrocardiography (to measure heart rate variability, HRV), and measure heart rate, blood pressure, lipids, HgbA1c, and inflammation/oxidation markers (leukocyte count, C-reactive protein, urinary F2 isoprostanes and exhaled nitric oxide). This research will show how product use-groups differ in response to acute product use and long-term use as they are related to key cardiovascular and pulmonary biomarkers. Objective measures of product use include exhaled CO and plasma nicotine/cotinine and urinary nicotine/cotinine concentrations. History of product use within use-groups will be related to biomarker status.

The proposed research will yield vital and comprehensive data regarding product use, subclinical arterial injury, atherosclerosis burden, arterial and pulmonary function, cardiac and aerobic fitness, cardiac autonomic regulation, systemic and pulmonary inflammation, and oxidative stress, as well as other key outcomes. These data will serve as a foundation for future longitudinal investigations of e-cigarette health effects and will inform public policy decisions, clinical intervention, and patient guidance regarding e-cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* able to read and write English
* no plans to quit smoking and/or e-cig use in the next month
* not using cigars/smokeless/snus tobacco >/= 1 time per week
* having a stable pattern of current product use
* able to walk at least 2 blocks without assistance or stopping
* Specific to Exclusive Smokers:

  * smokes daily
  * >/= 5 cigs/day for last 6 months
  * < 3 uses E-cigs in lifetime
  * >/= 5 ppm carbon monoxide (CO)
  * Cotinine > 100 ng/ml
* Specific to Exclusive E-cig users:

  * </= 2 days per month cigarette use for last 6 months
  * >/= 5 days per week E-cig use for last 3 months
  * </= 4 ppm CO
  * Cotinine > 100 ng/ml
* Specific to Never-users

  * < 100 cigarettes in a lifetime, none for > 5 years
  * < 3 E-cig uses in a lifetime
  * </= 4 ppm CO
  * Cotinine < 100 ng/ml

Exclusion Criteria:

* current use of a smoking cessation medication
* women who are pregnant or plan to get pregnant in the coming month
* women who might be pregnant
* incarcerated individuals
* history of sarcoidosis in past 5 years, or active interstitial lung/pulmonary fibrosis
* history of positive Coronavirus-19 test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 165 exclusive E-cig users, 165 exclusive cigarette smokers, and 110 never-users will be enrolled. Tobacco product use will be examined via time-line follow-back use-history measures, real-time measures, and lab measures. Potential participants will be assessed for eligibility via a phone screen. Because biomarker status may be affected by age and sex, groups will be stratified equally for gender (48/52 male/female) and age (≤35/>35 years).
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James H Stein, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Our plan includes the creation of a data archive with coded information in computer-readable form for distribution to the scientific community using the procedures outlined below. The information will include a codebook with definitions of variables, variable field locations, summary statistics and any standard scoring. Final data sets will be stripped of identifiers prior to release for sharing (the release of a limited data set containing one or more specific identifiers would be considered if absolutely required by the researcher and if the request meets all University of Wisconsin -Institutional Review Board and Office of Human Research Protections policies. We will make all key variables available via posting of final data codebook and dataset in suitable archives. All shared variables and datasets will be de-identified and approved for sharing by the University of Wisconsin and Institutional Review Board
Supporting Information: Study Protocol, SAP
Time Frame: After data has been collected and analyzed.
Access Criteria: In accord with an Institutional Review Board-approved study consent that will permit sharing of study data sets under University of Wisconsin and Institutional Review Board policies, University of Wisconsin Center for Tobacco Research and Intervention will act under its own auspices as the hub for making data related to these topics available. We will make the final de-identified study dataset available by request from other researchers in accord with NHLBI policy.
URL: http://www.ctri.wisc.edu

REFERENCES:
- [Result] Tattersall MC, Hughey CM, Piasecki TM, Korcarz CE, Hansen KM, Ott NR, Sandbo N, Fiore MC, Baker TB, Stein JH. Cardiovascular and Pulmonary Responses to Acute Use of Electronic Nicotine Delivery Systems and Combustible Cigarettes in Long-Term Users. Chest. 2023 Sep;164(3):757-769. doi: 10.1016/j.chest.2023.03.047. Epub 2023 Apr 10. PMID 37044158
- See also: link to full manuscript with published results for this trial — https://doi.org/10.1016/j.chest.2023.03.047

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 5 2019 started enrollment, ended last visit March 9th 2022. Studies were conducted at the University of Wisconsin Hospital and Clinics and the Center for Tobacco Research and Intervention (CTRI) in Madison, WI and for a short period we also at CTRI location in Milwaukee,WI.
Pre-assignment Details: Participants tested for Exhaled CO and urinary nicotine to determine if they qualified for either arm of the study. E-cigarette vapers exclusively (exhaled CO less than 5 ppm and nicotine in urine), cigarettes exclusively (CO more or equal 5 ppm, positive urine nicotine), and controls (CO less than 5 ppm, and negative nicotine in urine). NOTE: one participant was enrolled twice completing all study visits. Later, when this was noticed, we amended procedures, only his initial data was used.
Period: Overall Study
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Started | 139 | 192 | 119
Completed | 117 | 164 | 114
Not Completed | 22 | 28 | 5
Not completed — COVID-19 shutdown period | 0 | 4 | 0
Not completed — Missed V2 visit- outside protocol window | 4 | 3 | 1
Not completed — Lost to Follow-up | 8 | 0 | 2
Not completed — Did not qualify due to comorbidities, positive COVID-9, high CO, Low CO, Negative nicotine in urine | 10 | 20 | 2
Not completed — While cleaning datasets, we realized one participant was enrolled twice. | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: results are reported for only those participants who completed the final study visit, when outcome data was collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users | Total
Number analyzed (Participants) | 117 | 164 | 114 | 395
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (13.8) | 27.4 (10.6) | 30.8 (11.9) | 32.9 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 64 | 57 | 173
  Male | 65 | 100 | 57 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6 | 12
  Not Hispanic or Latino | 115 | 159 | 108 | 382
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 7 | 9 | 21 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 38 | 4 | 5 | 47
  White | 65 | 141 | 79 | 285
  More than one race | 5 | 9 | 9 | 23
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants] — 392 from Madison and 3 from Milwaukee, Wisconsin, USA
  participants
    United States | 117 | 164 | 114 | 395
Exhaled CO [Mean (Standard Deviation); unit: ppm] — Exhaled CO concentration at final visit after 8 hours refraining from smoking or vaping
  ppm | 16.11 (13.7) | 2.96 (1.89) | 2.79 (1.73) | 6.8 (9.7)
Serum Nicotine (ng/ml) [Mean (Standard Deviation); unit: ng/ml] — Serum Nicotine concentration at V2 after 8 hours of refraining from use of nicotine products.
  For these assays, the minimum value was coded as 1.99 when the concentration was below the threshold of detection (<2 ng/ml).
  ng/ml | 4.48 (4.54) | 2.95 (2.58) | 1.99 (0.00) | 3.07 (3.07)
Serum Cotinine (ng/ml) [Mean (Standard Deviation); unit: ng/ml] — Serum Cotinine concentration at V2 after 8 hours of refraining from use of nicotine products.
  For these assays, the minimum value was coded as 1.99 when the concentration was below the threshold of detection (<2 ng/ml).
  ng/ml | 231.3 (127.7) | 193.5 (111.7) | 2.99 (8.88) | 140.4 (141.0)

OUTCOME MEASURES:

1. Primary Outcome: Brachial Artery Flow-Mediated Dilation (FMD)- Pre Challenge
Description: Brachial Artery Flow-Mediated Dilation is a primary cardiovascular biomarker and a measure of endothelial function that will be assessed before and after an acute exposure challenge. These are pre-challenge values.
  Ultrasound based changes in brachial artery diameter after a forearm cuff occlusion (250mmHg) for 5 minutes. FMD is the percent change in brachial diameter measured 60 to 90 seconds post cuff release compared to its resting diameter. A higher % dilation is an indication of better endothelial function.
Time Frame: V2 up to 4 weeks from enrollment visit, fasting
Population: % FMD pre-challenge after 8 hours refraining from nicotine exposure. A higher % dilation is an indication of better endothelial function.
Measure: Mean (Standard Deviation); unit: Percent change from resting diameter
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Number analyzed (Participants) | 113 | 164 | 114
Percent change from resting diameter | 4.25 (3.17) | 4.89 (2.92) | 5.31 (3.43)
Statistical Analysis 1: Comparison: Exclusive Smokers vs Exclusive E-Cig Users vs Never Users; Test type: Other; p = .494, ANCOVA; Age, sex, and race/ethnicity were covaried. Test for group difference: F (2, 384) = 0.707, p = .494

2. Primary Outcome: Forced Expiratory Volume (FEV1)- Pre Challenge
Description: FEV1 is a primary measure of pulmonary disease obtained by spirometry that will be assessed before and after an acute exposure challenge. These are per-challenge values
Time Frame: V2 up to 4 weeks from enrollment visit , fasting, pre challenge session
Measure: Mean (Standard Deviation); unit: percentage of volume exhaled
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Number analyzed (Participants) | 112 | 162 | 114
percentage of volume exhaled | 82.9 (18.9) | 93.8 (13.3) | 92.0 (13.4)
Statistical Analysis 1: Comparison: Exclusive Smokers vs Exclusive E-Cig Users vs Never Users; Test type: Other; p = 0.001, ANCOVA; Age, sex, and race/ethnicity were covaried. Test for group difference F(2, 381) = 7.409, p = .001
Statistical Analysis 2: Comparison: Exclusive E-Cig Users vs Never Users; these are pairwise follow-up tests probing a larger omnibus group difference involving three groups; Test type: Other; p = 0.822, ANCOVA post-hoc pairwise group compariso; Age, sex, and race/ethnicity were covaried; Mean Difference (Final Values) = -0.420, 95% CI 2-sided [-4.080 to 3.240]
Statistical Analysis 3: Comparison: Exclusive Smokers vs Never Users; these are pairwise follow-up tests probing a larger omnibus group difference involving three groups; Test type: Other; p = 0.001, ANCOVA post-hoc pairwise group compariso; Age, sex, and race were covaried; Mean Difference (Final Values) = 7.267, 95% CI 2-sided [2.974 to 11.559]
Statistical Analysis 4: Comparison: Exclusive Smokers vs Exclusive E-Cig Users; These are pairwise follow-up tests probing a larger omnibus group difference involving three groups; Test type: Other; p < 0.001, ANCOVA post-hoc pairwise group compariso; Age, sex and race were covaried; Mean Difference (Final Values) = 7.687, 95% CI 2-sided [3.485 to 11.889]

3. Primary Outcome: Carotid Intima-Media Thickness (IMT)
Description: Carotid Intima-Media Thickness is a cardiovascular biomarker and a measure of sub-clinical arterial injury and atherosclerosis as a result of chronic exposure. IMT will be measured via ultrasonography.
Time Frame: V2 up to 4 weeks from enrollment visit, only done pre-challenge
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Number analyzed (Participants) | 116 | 164 | 113
mm | 0.67 (0.18) | 0.54 (0.10) | 0.54 (0.10)
Statistical Analysis 1: Comparison: Exclusive Smokers vs Exclusive E-Cig Users vs Never Users; Test type: Other; p = .074, ANCOVA — Age, sex, and race/ethnicity were covaried. Test for group difference: F (2, 386) = 2.616, p = .074

4. Primary Outcome: Changes in Systolic Blood Pressure Pre- and Post-challenge.
Description: Visit 2 was scheduled up to 4 weeks from enrollment visit, fasting.. They came in the morning after 8 hours of fasting and refraining from nicotine products. Systolic blood pressure (left brachial artery using an oscillometric method) was measured supine, after 10 minutes rest ("Pre") and repeated after they underwent smoking or vaping changes. The "post challenge" blood pressures were recorded 15-20 minutes post end of exposure. For controls, all measurements were repeated in the same order after a 10 minute break.
Time Frame: During Visit 2 (1 - 4 weeks post enrollment) before and after smoking/vaping challenge and for controls after a 10 minute break
Population: Not all controls (never users) were assessed post (after 10 minute break) due to time restrictions in personnel and one exclusive e-cigarette user was not assessed post due to a vaso-vagal response during blood draw.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Never Users - Pre: Control subjects at baseline
- Never Users-Post: Repeated assessment after 15 minutes of rest.
- Exclusive E-cigarette Users Pre Challenge: Electronic cigarette users assessed after 8 hours of refraining from vaping.
- Exclusive E-cigarette Users Post-challenge: Vapers completed a maximum of 15 minute ad libitum product use challenge , Vaping their own electronic cigarettes
- Exclusive Smokers Pre-challenge: Exclusive cigarette smokers assessed after 8 hours refraining from smoking
- Exclusive Smokers After Smoking Challenge: Smokers completed a maximum 15-minute ad libitum product use challenge, they smoked their combustible cigarettes in a dedicated room with external ventilation, under remote supervision by two trained observers.
Arm/Group | Never Users - Pre | Never Users-Post | Exclusive E-cigarette Users Pre Challenge | Exclusive E-cigarette Users Post-challenge | Exclusive Smokers Pre-challenge | Exclusive Smokers After Smoking Challenge
Number analyzed (Participants) | 114 | 99 | 164 | 163 | 115 | 115
mmHg | 118.4 (11.72) | 120.25 (12.00) | 119.74 (11.21) | 125.40 (11.54) | 126.43 (16.72) | 132.00 (16.09)
Statistical Analysis 1: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Linear mixed models adjusted for age, sex, race/ethnicity compared the within-and between-group responses following product use; Test type: Other; p = .002, Mixed Models Analysis — False Discovery Rate correction (Benjamini and Hochberg procedure) applied to a set of 13 Group x Time interaction tests; Omnibus Group x Time (pre-post) interaction test: F (2, 378.467) = 6.609, p = .002. Age, race, and sex were covaried; Type III F-test of Fixed Group x Time ef = 6.609 — F (2, 378.467) = 6.609, p = .002
Statistical Analysis 2: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge; Fixed effects from mixed models of measures before and after nicotine-containing product challenge (covariate-adjusted); Test type: Other; p = 0.001, Mixed Models Analysis; interaction estimate = 3.30, 95% CI 2-sided [1.36 to 5.24], Standard Error of Mean 0.99 — fixed effects from linear mixed model testing for effects of group, time, and group x time in systolic blood pressure, adjusting for age, sex, and race. Here presented the Exclusive E-cigarette users x Time vs never users x time as reference
Statistical Analysis 3: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.002, Mixed Models Analysis; interaction term estimate = 3.29, 95% CI 2-sided [1.20 to 5.38], Standard Error of Mean 1.06 — fixed effects from linear mixed model testing for effects of group, time, and group x time in systolic blood pressure, adjusting for age, sex, and race. Here presented the Exclusive cigarette smokers x Time vs never users x time as reference
Statistical Analysis 4: Comparison: Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = .992, ANCOVA; Mean Difference (Final Values) = 0.09, Standard Error of Mean 0.948

5. Primary Outcome: Changes in Diastolic Blood Pressure Pre- and Post-challenge.
Description: Participants returned for V2 up to 4 weeks from enrollment visit, fasting. They came in the morning after 8 hours of fasting and refraining from nicotine products. Diastolic blood pressure (left brachial artery using an oscillometric method) was measured supine, after 10 minutes rest ("Pre") and repeated after they underwent smoking or vaping changes. The "post challenge" blood pressures were recorded 15-20 minutes post end of exposure. For controls, all measurements were repeated in the same order after a 10 minute break.
Time Frame: before and after smoking/vaping challenge during Visit 2 (up to 4 weeks from enrollment)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Never Users - Pre | Never Users-Post | Exclusive E-cigarette Users Pre Challenge | Exclusive E-cigarette Users Post-challenge | Exclusive Smokers Pre-challenge | Exclusive Smokers After Smoking Challenge
Number analyzed (Participants) | 114 | 99 | 164 | 163 | 115 | 115
mmHg | 70.40 (7.13) | 72.51 (7.73) | 71.12 (7.52) | 75.31 (8.54) | 76.64 (10.72) | 81.04 (10.78)
Statistical Analysis 1: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.003, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Age, race, and sex were covaried. Omnibus Group x Time (pre-post) interaction test: F (2, 378.999) = 5.843, p = .003; Type III F-test of Fixed Group x Time ef = 5.843 — F (2, 378.999) = 5.843, p = .003
Statistical Analysis 2: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge; Fixed effects from mixed models of measures before and after nicotine-containing product challenge (covariate-adjusted); Test type: Other; p = .002, Mixed Models Analysis; Interaction term Coefficient = 0.03, 95% CI 2-sided [0.01 to 0.05], Standard Error of Mean 0.01 — fixed effects from linear mixed model testing for effects of group, time, and group x time in diastolic blood pressure, adjusting for age, sex, and race. Here presented the Exclusive E-cigarette users x Time vs never users x time as reference
Statistical Analysis 3: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Fixed effects from mixed models of measures before and after nicotine-containing product challenge (covariate-adjusted); Test type: Other; p = .003, Mixed Models Analysis; Interaction term Coefficient = 0.03, 95% CI 2-sided [0.01 to 0.05], Standard Error of Mean 0.01 — fixed effects from linear mixed model testing for effects of group, time, and group x time in diastolic blood pressure, adjusting for age, sex, and race. Here presented the Exclusive Smokers x Time vs never users x time as reference
Statistical Analysis 4: Comparison: Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Fixed effects from mixed models of measures before and after nicotine-containing product challenge (covariate-adjusted); Test type: Other; p = .917, Mixed Models Analysis; Interaction term Coefficient = 0.00, Standard Error of Mean 0.01 — fixed effects from re-parameterized linear mixed model testing for effects of group, time, and group x time in diastolic blood pressure, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs Exclusive Smokers x time as reference

6. Primary Outcome: Changes in Heart Rate Pre- and Post-challenge.
Description: Visit 2 was scheduled up to 4 weeks from enrollment visit, fasting. Participants attended fasting and refraining from nicotine products for at least 8 hours prior. All visits were in the morning. Pre-challenge heart rate measured supine, after 10 minutes rest from blood pressure monitor (dinamap). The post challenge heart rates were recorded 15-20 minutes post end of exposure to smoking or vaping challenge completion or in the case of controls after a 10 minute break.
Time Frame: Before and after smoking/vaping challenge during Visit 2 (up to 4 weeks from enrollment)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Never Users - Pre | Never Users-Post | Exclusive E-cigarette Users Pre Challenge | Exclusive E-cigarette Users Post-challenge | Exclusive Smokers Pre-challenge | Exclusive Smokers After Smoking Challenge
Number analyzed (Participants) | 114 | 99 | 164 | 163 | 115 | 115
beats per minute (bpm) | 59.57 (8.19) | 58.42 (7.88) | 58.34 (9.22) | 63.17 (10.13) | 65.31 (11.65) | 69.15 (12.05)
Statistical Analysis 1: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; [analysis description as in outcome 4, analysis 1]; Test type: Other; p < .001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Age, race, and sex were covaried. Omnibus Group x Time (pre-post) interaction test: F (2, 376.099) = 49.420, p < .001; Type III F-test of Fixed Group x Time Ef = 49.42 — F (2, 376.099) = 49.420, p < .001
Statistical Analysis 2: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge; Fixed effects from mixed models of measures before and after nicotine-containing product challenge (covariate-adjusted); Test type: Other; p < 0.001, Mixed Models Analysis; interaction term coefficient = 6.06, 95% CI 2-sided [4.83 to 7.3], Standard Error of Mean 0.63 — fixed effects from linear mixed model testing for effects of group, time, and group x time in Heart Rate, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs never users x time as reference
Statistical Analysis 3: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p < 0.001, Mixed Models Analysis; interaction term coefficient = 5.09, 95% CI 2-sided [3.76 to 6.42], Standard Error of Mean 0.68 — fixed effects from linear mixed model testing for effects of group, time, and group x time in Heart Rate, adjusting for age, sex, and race for Exclusive Smokers x Time vs never users x time as reference
Statistical Analysis 4: Comparison: Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.107, Mixed Models Analysis; interaction term coefficient = -0.97, Standard Error of Mean 0.602 — fixed effects from re-parameterized linear mixed model testing for effects of group, time, and group x time in Heart Rate, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs Exclusive Smokers x time as reference

7. Primary Outcome: Changes in Brachial Artery Diameter Pre- and Post-challenge
Description: Visit 2 was scheduled up to 4 weeks from enrollment visit. Participants attended fasting and refraining from nicotine products for at least 8 hours prior. All visits were in the morning. Pre-challenge brachial artery diameter imaged with ultrasound after resting supine for 10 minutes before and repeated 15-20 minutes after smoking/vaping challenge ended. or in the case of controls after a 10 minute break.
Time Frame: before and after smoking/vaping challenge during Visit 2 (up to 4 weeks from enrollment)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Never Users - Pre | Never Users-Post | Exclusive E-cigarette Users Pre Challenge | Exclusive E-cigarette Users Post-challenge | Exclusive Smokers Pre-challenge | Exclusive Smokers After Smoking Challenge
Number analyzed (Participants) | 114 | 99 | 164 | 163 | 113 | 113
centimeters (cm) | 0.378 (0.062) | 0.370 (0.063) | 0.388 (0.064) | 0.378 (0.063) | 0.410 (0073) | 0.398 (0.068)
Statistical Analysis 1: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.002, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Age, race, and sex were covaried. Omnibus Group x Time (pre-post) interaction test: F (2,372.971) = 6.194, p = .002; Type III F-test of Fixed Group x Time Ef = 6.194 — F (2,372.971) = 6.194, p = .002
Statistical Analysis 2: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge; Fixed effects from mixed models of measures before and after nicotine-containing product challenge (covariate-adjusted); Test type: Other; p = 0.003, Mixed Models Analysis; interaction term coefficient = -0.005, 95% CI 2-sided [-0.01 to -0.002], Standard Error of Mean 0.001 — fixed effects from linear mixed model testing for effects of group, time, and group x time in Brachial Artery Diameter, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs never users x time as reference
Statistical Analysis 3: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.001, Mixed Models Analysis; interaction term coefficient = -0.01, 95% CI 2-sided [-0.01 to -0.002], Standard Error of Mean 0.002 — fixed effects from linear mixed model testing for effects of group, time, and group x time in Brachial Artery Diameter, adjusting for age, sex, and race for Exclusive Smokers x Time vs never users x time as reference
Statistical Analysis 4: Comparison: Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.582, Mixed Models Analysis; interaction term coefficient = -0.001, Standard Error of Mean 0.002 — fixed effects from re-parameterized linear mixed model testing for effects of group, time, and group x time in Brachial Artery Diameter, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs Exclusive Smokers x time as reference

8. Primary Outcome: Changes in Brachial Artery Flow Mediated Dilation (FMD) Pre- and Post-challenge
Description: Visit 2 was scheduled up to 4 weeks from enrollment visit. Participants attended fasting and refraining from nicotine products for at least 8 hours prior. All visits were in the morning. Pre-challenge ultrasound of brachial artery diameter imaged with ultrasound after resting supine for 10 minutes before and repeated 15-20 minutes after smoking/vaping challenge ended. or in the case of controls after a 10 minute break. The FMD protocol includes measuring % change in resting diameter after 60-90 seconds post fore-arm cuff occlusion release.
Time Frame: Testing was done after 10 minutes rest and fasting for pre- and post-challenge. The post challenge FMD were recorded 15-20 minuted after end of exposure (up to 4 weeks from enrollment)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Never Users - Pre | Never Users-Post | Exclusive E-cigarette Users Pre Challenge | Exclusive E-cigarette Users Post-challenge | Exclusive Smokers Pre-challenge | Exclusive Smokers After Smoking Challenge
Number analyzed (Participants) | 114 | 99 | 164 | 163 | 113 | 113
percent change | 5.31 (3.43) | 4.22 (3.01) | 4.89 (2.92) | 4.62 (3.52) | 4.25 (3.17) | 3.57 (2.26)
Statistical Analysis 1: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.175, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Age, race, and sex were covaried; Type III F-test of Fixed Group x Time E = 1.753 — FMD responses in e-cigarette users, cigarette users, and never-users controls after adjusting for changes in brachial artery diameter
Statistical Analysis 2: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge; Fixed effects from mixed models of measures before and after nicotine-containing product challenge (covariate-adjusted); Test type: Other; p = 0.067, Mixed Models Analysis; interaction term coefficient = 0.75, 95% CI 2-sided [-0.05 to 1.56], Standard Error of Mean 0.41 — fixed effects from linear mixed model testing for effects of group, time, and group x time in Brachial Artery Flow Mediated Dilation, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs never users x time as reference
Statistical Analysis 3: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.464, Mixed Models Analysis; interaction term coefficient = 0.33, 95% CI 2-sided [-0.55 to 1.20], Standard Error of Mean 0.44 — fixed effects from linear mixed model testing for effects of group, time, and group x time in Brachial Artery Flow Mediated Dilation, adjusting for age, sex, and race for Exclusive Smokers x Time vs never users x time as reference
Statistical Analysis 4: Comparison: Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.284, Mixed Models Analysis; interaction term coefficient = -0.43, Standard Error of Mean 0.4 — fixed effects from re-parameterized linear mixed model testing effects of group, time, and group x time in FMD, age, sex, race adjusted, for Exclusive E-cigarette users x Time vs Exclusive Smokers x time as reference

9. Primary Outcome: Changes in Percent of Sequential Heart Cycles That Differ by More Than 50 ms From Each Other in Length (PNN50, %) Pre- and Post-challenge
Description: Expressed as a percentage of beats (supine recordings had be 5 minutes or longer to be valid). We used the SphygmoCor system for these recordings (Atcor medical). Participants attended V2 1-2 weeks after enrollment visit. They came in the morning fasting and refraining from nicotine for at least 8 hours. Heart rate variability was recorded supine for 10 minutes or more, pre and post smoking/vaping challenge. For controls is was repeated after a 10-minute break.
Time Frame: During V2 (scheduled up to 4 weeks from enrollment) and obtained after 10 minutes of supine rest, before and after smoking/vaping challenge
Population: Not all controls (never users) were assessed post (after 10 minute break) due to time restrictions in personnel and one exclusive e-cigarette user was not assessed post due to a vaso-vagal response during blood draw. Some participants pre or post challenge due to poor ECG signals (noise) or frequent premature ventricular contractions did not have a usable 10 minute recording
Measure: Mean (Standard Deviation); unit: percent of sequential intervals
Arm/Group | Never Users - Pre | Never Users-Post | Exclusive E-cigarette Users Pre Challenge | Exclusive E-cigarette Users Post-challenge | Exclusive Smokers Pre-challenge | Exclusive Smokers After Smoking Challenge
Number analyzed (Participants) | 105 | 92 | 158 | 152 | 105 | 110
percent of sequential intervals | 33.64 (20.83) | 36.46 (21.96) | 34.82 (21.85) | 31.02 (22.90) | 18.46 (19.72) | 15.45 (18.61)
Statistical Analysis 1: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; [analysis description as in outcome 4, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Age, race, and sex were covaried. Omnibus Group x Time (pre-post) interaction test: F (2, 342.847) = 8.323, p = <.001; Type III F-test of Fixed Group x Time Ef = 8.323 — F (2,342.847) = 8.323, p = <.001
Statistical Analysis 2: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge; Fixed effects from mixed models of measures before and after nicotine-containing product challenge (covariate-adjusted); Test type: Other; p < 0.001, Mixed Models Analysis; interaction term coefficient = -6.55, 95% CI 2-sided [-9.89 to -3.20], Standard Error of Mean 1.7 — fixed effects from linear mixed model testing for effects of group, time, and group x time in PNN50, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs never users x time as reference
Statistical Analysis 3: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.001, Mixed Models Analysis; interaction term coefficient = -6.11, 95% CI 2-sided [-9.71 to -2.52], Standard Error of Mean 1.83 — fixed effects from linear mixed model testing for effects of group, time, and group x time in PNN50, adjusting for age, sex, and race for Exclusive Smokers x Time vs never users x time as reference
Statistical Analysis 4: Comparison: Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.787, Mixed Models Analysis; interaction term coefficient = 0.44, Standard Error of Mean 1.61 — fixed effects from re-parameterized linear mixed model testing for effects of group, time, and group x time in PNN50, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs Exclusive Smokers x time as reference

10. Primary Outcome: Changes in Root Mean Square of Successive Differences Between Normal Heart Beats (RMSSD, ms) Pre- and Post-challenge
Description: Participants attended V2 up to 4 weeks after enrollment visit. They came in the morning fasting and refraining from nicotine for at least 8 hours. Heart rate variability was recorded supine for 10 minutes or more, pre and post smoking/vaping challenge. For controls it was repeated after a 10 minute break.
Time Frame: heart rate variability recordings of at least 10 minutes per-challenge and 15 minutes post-challenge (up to 4 weeks from enrollment)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Never Users - Pre | Never Users-Post | Exclusive E-cigarette Users Pre Challenge | Exclusive E-cigarette Users Post-challenge | Exclusive Smokers Pre-challenge | Exclusive Smokers After Smoking Challenge
Number analyzed (Participants) | 105 | 92 | 158 | 152 | 105 | 110
milliseconds | 66.44 (34.49) | 71.10 (38.78) | 71.20 (44.42) | 64.40 (46.33) | 48.29 (35.01) | 44.44 (38.73)
Statistical Analysis 1: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Linear mixed models adjusted for age, sex, race/ethnicity compared the within-and between-group responses following product use Outcome measure ln transformed for analysis; Test type: Other; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Age, race, and sex were covaried. Omnibus Group x Time (pre-post) interaction test: F (2, 345.918) = 7.260, p = .001; Type III F-test of Fixed Group x Time Ef = 7.26 — F (2,345.918) = 7.260, p = .001
Statistical Analysis 2: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge; Fixed effects from mixed models of measures before and after nicotine-containing product challenge (covariate-adjusted); Test type: Other; p = 0.001, Mixed Models Analysis; interaction term coefficient = -0.2, 95% CI 2-sided [-0.31 to -0.08], Standard Error of Mean 0.06 — fixed effects from linear mixed model testing for effects of group, time, and group x time in RMSSD, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs never users x time as reference
Statistical Analysis 3: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.001, Mixed Models Analysis; interaction term coefficient = -0.21, 95% CI 2-sided [-0.33 to -0.09], Standard Error of Mean 0.06 — fixed effects from linear mixed model testing for effects of group, time, and group x time in RMSSD, adjusting for age, sex, and race for Exclusive Smokers x Time vs never users x time as reference
Statistical Analysis 4: Comparison: Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.847, Mixed Models Analysis; interaction term coefficient = -0.01, Standard Error of Mean 0.05 — fixed effects from re-parameterized linear mixed model testing for effects of group, time, and group x time in RMSSD, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs Exclusive Smokers x time as reference

11. Primary Outcome: Changes in Heart Rate Variability Standing Ratio Pre- and Postchallenge
Description: We used the SphygmoCor system for these recordings (Atcor medical). Participants attended V2 up to 4 weeks after enrollment visit. They came in the morning fasting and refraining from nicotine for at least 8 hours. Heart rate variability standing ratio was assessed pre and post smoking/vaping challenge. For controls is was repeated after a 10-minute break. Ratio between maximal heart rate after abrupt standing from a supine position and the subsequent lowest heart rate value within 40 seconds of peak.
Time Frame: Ratio was measured pre- and post- smoking/vaping challenge after completion of the 10 minutes of heart rate variability measures (up to 4 weeks from enrollment)
Population: Not all controls (never users) were assessed post (after 10 minute break) due to time restrictions in personnel and one exclusive e-cigarette user was not assessed post due to a vaso-vagal response during blood draw. Some participants pre or post challenge due to poor ECG signals (noise) or frequent premature ventricular contractions did not have a usable recording
Measure: Mean (Standard Deviation); unit: ratio (unitless)
Arm/Group | Never Users - Pre | Never Users-Post | Exclusive E-cigarette Users Pre Challenge | Exclusive E-cigarette Users Post-challenge | Exclusive Smokers Pre-challenge | Exclusive Smokers After Smoking Challenge
Number analyzed (Participants) | 105 | 85 | 139 | 140 | 94 | 84
ratio (unitless) | 1.57 (0.26) | 1.55 (0.22) | 1.55 (0.23) | 1.51 (0.23) | 1.38 (0.21) | 1.34 (0.23)
Statistical Analysis 1: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = .182, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Age, race, and sex were covaried. Omnibus Group x Time (pre-post) interaction test: F (2, 312.081) = 1.712, p = .182; Type III F-test of Fixed Group x Time Ef = 1.712 — F (2, 312.081) = 1.712, p = .182
Statistical Analysis 2: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge; Test type: Other; p = 0.07, Mixed Models Analysis; interaction term coefficient = -0.04, 95% CI 2-sided [-0.09 to 0.004], Standard Error of Mean 0.02 — fixed effects from linear mixed model testing for effects of group, time, and group x time in HRV-Standing Ratio, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs never users x time as reference
Statistical Analysis 3: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.196, Mixed Models Analysis; interaction term coefficient = -0.03, 95% CI 2-sided [-0.09 to 0.02], Standard Error of Mean 0.03 — fixed effects from linear mixed model testing for effects of group, time, and group x time in HRV-Standing Ratio adjusting for age, sex, and race for Exclusive Smokers x Time vs never users x time as reference
Statistical Analysis 4: Comparison: Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.69, Mixed Models Analysis; interaction term coefficient = 0.09, Standard Error of Mean 0.02 — fixed effects from re-parameterized linear mixed model testing for effects of group, time, and group x time in HRV-Standing Ratio adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs Exclusive Smokers x time as reference

12. Primary Outcome: Changes in Predicted Forced Expiatory Volume in 1 Second (FEV1, %) Pre- and Post-challenge
Description: maximum amount of air that the subject can forcibly expel during the first second following maximal inhalation, expressed as a percentage of the predicted normal values in the population. Participants attended V2 1-4 weeks after enrollment. They came in the morning, fasting and refraining from nicotine exposure for at least 8 hours prior. Pre-challenge spirometry was performed sitting before all other tests and repeated within 15 minutes after smoking/vaping challenge.
Time Frame: before and after smoking/vaping challenge during Visit 2 (1-4 weeks after enrollment visit)
Population: Not all controls (never users) were assessed post (after 10 minute break) due to time restrictions in personnel and one exclusive e-cigarette user was not assessed post due to a vaso-vagal response during blood draw. Some spirometry recordings were of poor quality and upon review by pulmonologist they were deemed not usable.
Measure: Mean (Standard Deviation); unit: predicted percentage of population
Arm/Group | Never Users - Pre | Never Users-Post | Exclusive E-cigarette Users Pre Challenge | Exclusive E-cigarette Users Post-challenge | Exclusive Smokers Pre-challenge | Exclusive Smokers After Smoking Challenge
Number analyzed (Participants) | 114 | 100 | 162 | 161 | 112 | 111
predicted percentage of population | 92.00 (13.41) | 91.12 (14.13) | 93.83 (13.32) | 89.76 (15.63) | 82.91 (18.90) | 80.43 (18.25)
Statistical Analysis 1: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.017, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Age, race, and sex were covaried. Omnibus Group x Time (pre-post) interaction test: F (2, 373.239) = 4.096, p = .017; Type III F-test of Fixed Group x Time Ef = 4.096 — F (2, 373.239) = 4.096, p = .017
Statistical Analysis 2: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge; Test type: Other; p = 0.005, Mixed Models Analysis; interaction term coefficient = -3.04, 95% CI 2-sided [-5.18 to -0.91], Standard Error of Mean 1.09 — fixed effects from linear mixed model testing for effects of group, time, and group x time in FEV1, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs never users x time as reference
Statistical Analysis 3: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.274, Mixed Models Analysis; interaction term coefficient = -1.29, 95% CI 2-sided [-3.61 to 1.03], Standard Error of Mean 1.18 — fixed effects from linear mixed model testing for effects of group, time, and group x time in FEV1, adjusting for age, sex, and race for Exclusive Smokers x Time vs never users x time as reference
Statistical Analysis 4: Comparison: Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.098, Mixed Models Analysis; interaction term coefficient = 1.75, Standard Error of Mean 1.06 — fixed effects from re-parameterized linear mixed model testing for effects of group, time, and group x time in FEV1, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs Exclusive Smokers x time as reference

13. Primary Outcome: Changes in Forced Vital Capacity (FVC, %) Pre- and Post-Challenge.
Description: Amount of air that can be forcibly exhaled after taking the deepest breath possible expressed as a predicted percentage from the normal population. Participants attended V2 1-4 weeks after enrollment. They came in the morning, fasting and refraining from nicotine exposure for at least 8 hours prior. Pre-challenge spirometry was performed sitting before all other tests and repeated within 15 minutes after smoking/vaping challenge.
Time Frame: before and after smoking/vaping challenge during Visit 2 Visit 2 which was scheduled 1 to 4 weeks from enrollment visit, fasting
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: predicted percentile
Arm/Group | Never Users - Pre | Never Users-Post | Exclusive E-cigarette Users Pre Challenge | Exclusive E-cigarette Users Post-challenge | Exclusive Smokers Pre-challenge | Exclusive Smokers After Smoking Challenge
Number analyzed (Participants) | 114 | 100 | 162 | 161 | 112 | 111
predicted percentile | 96.45 (15.06) | 95.00 (14.19) | 98.25 (13.50) | 96.77 (15.79) | 90.28 (15.99) | 87.88 (16.55)
Statistical Analysis 1: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = .771, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Age, race, and sex were covaried. Omnibus Group x Time (pre-post) interaction test: F (2, 373.434) = 0.260, p = .771; Type III F-test of Fixed Group x Time Ef = 0.26 — F (2, 373.434) = 0.260, p = .771
Statistical Analysis 2: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge; Fixed effects from mixed models of measures before and after nicotine-containing product challenge (covariate-adjusted); Test type: Other; p = 0.918, Mixed Models Analysis; interaction term coefficient = -0.12, 95% CI 2-sided [-2.35 to 2.12], Standard Error of Mean 1.14 — fixed effects from linear mixed model testing for effects of group, time, and group x time in FVC, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs never users x time as reference
Statistical Analysis 3: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.518, Mixed Models Analysis; interaction term coefficient = -0.8, 95% CI 2-sided [-3.22 to 1.63], Standard Error of Mean 1.23 — fixed effects from linear mixed model testing for effects of group, time, and group x time in FVC, adjusting for age, sex, and race for Exclusive Smokers x Time vs never users x time as reference
Statistical Analysis 4: Comparison: Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.539, Mixed Models Analysis; interaction term coefficient = -0.68, Standard Error of Mean 1.11 — fixed effects from re-parameterized linear mixed model testing for effects of group, time, and group x time in FVC, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs Exclusive Smokers x time as reference

14. Primary Outcome: Changes in Ratio Between Predicted Forced Expiatory Volume in First Second and Predicted Total Vital Capacity (FEV1/FVC Ratio) Pre- and Post-challenge
Description: The post challenge spirometry was recorded <15 minutes post end of exposure. Participants attended V2 1-4 weeks after enrollment. They came in the morning, fasting and refraining from nicotine exposure for at least 8 hours prior. Pre-challenge spirometry was performed sitting before all other tests and repeated within 15 minutes after smoking/vaping challenge.
Time Frame: before and after smoking/vaping challenge during Visit 2 (1-4 weeks after enrollment visit)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ratio (unitless)
Arm/Group | Never Users - Pre | Never Users-Post | Exclusive E-cigarette Users Pre Challenge | Exclusive E-cigarette Users Post-challenge | Exclusive Smokers Pre-challenge | Exclusive Smokers After Smoking Challenge
Number analyzed (Participants) | 114 | 100 | 162 | 161 | 112 | 111
ratio (unitless) | 95.74 (9.63) | 95.93 (8.28) | 95.66 (8.90) | 92.23 (11.67) | 91.18 (12.56) | 90.89 (11.12)
Statistical Analysis 1: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Age, race, and sex were covaried. Omnibus Group x Time (pre-post) interaction test: F (2, 375.412) = 7.157, p = .001; Type III F-test of Fixed Group x Time Ef = 7.157 — F (2, 375.412) = 7.157, p = .001
Statistical Analysis 2: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge; Test type: Other; p = 0.001, Mixed Models Analysis; interaction term coefficient = -3.39, 95% CI 2-sided [-5.43 to -1.35], Standard Error of Mean 1.04 — fixed effects from linear mixed model testing for effects of group, time, and group x time in FEV1/FVC, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs never users x time as reference
Statistical Analysis 3: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.778, Mixed Models Analysis; interaction term coefficient = -0.32, 95% CI 2-sided [-2.53 to 1.89], Standard Error of Mean 1.12 — fixed effects from linear mixed model testing for effects of group, time, and group x time in FEV1/FVC, adjusting for age, sex, and race for Exclusive Smokers x Time vs never users x time as reference
Statistical Analysis 4: Comparison: Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.002, Mixed Models Analysis; interaction term coefficient = 3.08, Standard Error of Mean 1.08 — fixed effects from re-parameterized linear mixed model testing for effects of group, time, and group x time in FEV1/FVC, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs Exclusive Smokers x time as reference

15. Primary Outcome: Changes in Percent Predicted Forced Expiratory Flow at 25 and 75% of the Pulmonary Volume (FEF 25-75, %) Pre and Pos-challenge
Description: Participants attended Visit 2 (1-4 weeks after enrollment visit). They came in the morning, fasting and refraining from nicotine exposure for at least 8 hours prior. Pre-challenge spirometry was performed sitting before all other tests and repeated within 15 minutes after smoking/vaping challenge.
Time Frame: Spirometry performed pre-challenge and within 15 minutes post-challenge (up to 4 weeks from enrollment)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: predicted percentile
Arm/Group | Never Users - Pre | Never Users-Post | Exclusive E-cigarette Users Pre Challenge | Exclusive E-cigarette Users Post-challenge | Exclusive Smokers Pre-challenge | Exclusive Smokers After Smoking Challenge
Number analyzed (Participants) | 114 | 100 | 162 | 161 | 112 | 111
predicted percentile | 86.91 (27.33) | 85.17 (25.68) | 87.94 (23.45) | 80.20 (23.35) | 71.09 (31.09) | 68.49 (27.12)
Statistical Analysis 1: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.014, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Age, race, and sex were covaried. Omnibus Group x Time (pre-post) interaction test: F (2, 373.170) = 4.317, p = .014; Type III F-test of Fixed Group x Time Ef = 4.317 — F (2, 373.170) = 4.317, p = .014
Statistical Analysis 2: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge; Fixed effects from mixed models of measures before and after nicotine-containing product challenge (covariate-adjusted); Test type: Other; p = 0.016, Mixed Models Analysis; interaction term coefficient = -5.08, 95% CI 2-sided [-9.21 to -0.95], Standard Error of Mean 2.1 — fixed effects from linear mixed model testing for effects of group, time, and group x time in FEF 25-75, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs never users x time as reference
Statistical Analysis 3: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.998, Mixed Models Analysis; interaction term coefficient = 0.01, 95% CI 2-sided [-4.47 to 4.48], Standard Error of Mean 2.28 — fixed effects from linear mixed model testing for effects of group, time, and group x time in FEF 25-75, adjusting for age, sex, and race for Exclusive Smokers x Time vs never users x time as reference
Statistical Analysis 4: Comparison: Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.013, Mixed Models Analysis; interaction term coefficient = 5.09, Standard Error of Mean 2.04 — fixed effects from re-parameterized linear mixed model testing for effects of group, time, and group x time in FEF 25-75, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs Exclusive Smokers x time as reference

16. Primary Outcome: Changes in Fractional Exhaled Nitric Oxide (FeNO, Ppb) Pre- and Post-challenge
Description: Participants attended V2 1-4 weeks after enrollment. They came in the morning, fasting and refraining from nicotine exposure for at least 8 hours prior. Pre-challenge FeNO was obtained sitting and repeated within 15 minutes after smoking/vaping challenge.
Time Frame: before and after less than 15 minutes from smoking/ vaping product (up to 4 weeks from enrollment)
Population: Not all controls (never users) were assessed post (after 10 minute break) due to time restrictions in personnel and one exclusive e-cigarette user was not assessed post due to a vaso-vagal response during blood draw. Other missing records were due to equipment malfunction or participant not being able to follow instructions to complete the test correctly.
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Arm/Group | Never Users - Pre | Never Users-Post | Exclusive E-cigarette Users Pre Challenge | Exclusive E-cigarette Users Post-challenge | Exclusive Smokers Pre-challenge | Exclusive Smokers After Smoking Challenge
Number analyzed (Participants) | 114 | 100 | 163 | 161 | 111 | 108
parts per billion (ppb) | 16.17 (11.04) | 16.97 (12.52) | 14.51 (14.71) | 13.64 (14.47) | 9.67 (12.26) | 9.93 (11.84)
Statistical Analysis 1: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Linear mixed models adjusted for age, sex, race/ethnicity compared the within-and-between-group responses following product use Outcome measure ln transformed for analysis; Test type: Other; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Age, race, and sex were covaried. Omnibus Group x Time (pre-post) interaction test: F (2,376.779) = 6.694, p = .001; Type III F-test of Fixed Group x Time Ef = 6.694 — F ((2,376.779) = 6.694, p = .001
Statistical Analysis 2: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge; Fixed effects from mixed models of measures before and after nicotine-containing product challenge (covariate-adjusted); Test type: Other; p = 0.001, Mixed Models Analysis; interaction term coefficient = -0.09, 95% CI 2-sided [-0.14 to -0.04], Standard Error of Mean 0.03 — fixed effects from linear mixed model testing for effects of group, time, and group x time in FeNO, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs never users x time as reference
Statistical Analysis 3: Comparison: Never Users - Pre vs Never Users-Post vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.555, Mixed Models Analysis; interaction term coefficient = -0.02, 95% CI 2-sided [-0.08 to 0.04], Standard Error of Mean 0.03 — fixed effects from linear mixed model testing for effects of group, time, and group x time in FeNO, adjusting for age, sex, and race for Exclusive Smokers x Time vs never users x time as reference
Statistical Analysis 4: Comparison: Exclusive E-cigarette Users Pre Challenge vs Exclusive E-cigarette Users Post-challenge vs Exclusive Smokers Pre-challenge vs Exclusive Smokers After Smoking Challenge; Test type: Other; p = 0.007, Mixed Models Analysis; interaction term coefficient = 0.007, Standard Error of Mean 0.03 — fixed effects from re-parameterized linear mixed model testing for effects of group, time, and group x time in FeNO, adjusting for age, sex, and race for Exclusive E-cigarette users x Time vs Exclusive Smokers x time as reference

17. Secondary Outcome: Heart Rate (HR)
Description: Heart Rate pre-acute exposure challenge was obtained after resting supine for 10 minutes during V2 in the morning, fasting and refraining from nicotine exposure for at least 8 hours prior.
Time Frame: Participants attended V2 generally 1-4 weeks after enrollment with a window that allowed up to 4 weeks after enrollment
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Number analyzed (Participants) | 115 | 164 | 114
beats/minute | 65.3 (11.7) | 58.3 (9.2) | 59.6 (8.2)
Statistical Analysis 1: Comparison: Exclusive Smokers vs Exclusive E-Cig Users vs Never Users; Test type: Other; p < .001, ANCOVA — ANCOVA for group differences; Age, sex, and race/ethnicity were covaried. Test for group difference: F (2, 386) = 12.869, p < .001
Statistical Analysis 2: Comparison: Exclusive E-Cig Users vs Never Users; Never Users minus Exclusive E-Cig Users; Test type: Other; p = 0.269, ANCOVA post-hoc pairwise group compariso; Age, sex, and race were covaried; Mean Difference (Final Values) = 1.352, 95% CI 2-sided [-1.048 to 3.752]
Statistical Analysis 3: Comparison: Exclusive Smokers vs Never Users; Never Users minus Exclusive Smokers; Test type: Other; p < 0.001, ANCOVA post-hoc pairwise group compariso; Age, sex and race were covaried; Mean Difference (Final Values) = -5.575, 95% CI 2-sided [-8.37 to -2.780]
Statistical Analysis 4: Comparison: Exclusive Smokers vs Exclusive E-Cig Users; Exclusive E-Cig Users minus Exclusive Smokers; Test type: Other; p < 0.001, ANCOVA post-hoc pairwise group compariso; Age, sex and race were covaried; Mean Difference (Final Values) = -6.927, 95% CI 2-sided [-9.672 to -4.183]

18. Secondary Outcome: Heart Rate Variability (HRV) - Pre Product Use Challenge
Description: Heart Rate Variability PNN50(%) measured before an exposure challenge. Participants attended visit 2 fasting and refraining from nicotine for at least 8 hours.
Time Frame: V2 two was generally scheduled 1-4 weeks after enrollment visit with a window up to 4 weeks. HRV measures obtained after resting supine for 10 minutes
Population: heart rate variability depends on a good quality electrocardiogram, and some participants due to noise, significant pauses, very slow heart rate or frequent premature ventricular contractions did not have usable records, hence lower number analyzed.
Measure: Median (Inter-Quartile Range); unit: percentage of intervals
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Number analyzed (Participants) | 105 | 158 | 105
percentage of intervals | 11.4 [2.3 to 27.95] | 37.1 [15.0 to 51.98] | 31.0 [16.05 to 48.80]
Statistical Analysis 1: Comparison: Exclusive Smokers vs Exclusive E-Cig Users vs Never Users; Test type: Other; p = .035, ANCOVA; Age, sex, and race/ethnicity were covaried. Test for group difference: F (2, 361) = 3.392, p = .035; Group difference did not survive correction for false discovery rate at .05, therefore not followed with post-hoc pairwise comparisons

19. Secondary Outcome: Systolic Blood Pressure (BP)
Description: Blood Pressure measured using the oscillometric technique before an acute exposure challenge following standardized protocol. After resting supine for 10 minutes blood pressure was measured on both arms and the average of the last two values was used.
Time Frame: V2 was up to 4 weeks from enrollment visit, after resting supine for 10 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Number analyzed (Participants) | 115 | 164 | 114
mmHg | 126.4 (16.7) | 119.7 (11.2) | 118.4 (11.7)
Statistical Analysis 1: Comparison: Exclusive Smokers vs Exclusive E-Cig Users vs Never Users; Test type: Other; p = .549, ANCOVA; Age, sex, and race/ethnicity were covaried. Test for group difference: F (2, 386) = 0.601, p = .549

20. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Forced Vital Capacity is a measure of how much air can be exhaled forcefully obtained by spirometry pre acute exposure challenge.
Time Frame: recordings obtained during V2 in the morning, fasting and refraining from nicotine for at least 8 hours. This visit was generally 1-2 weeks after enrollment date with a window up to 4 weeks
Measure: Mean (Standard Deviation); unit: Percent predicted FVC
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Number analyzed (Participants) | 112 | 162 | 114
Percent predicted FVC | 90.3 (16) | 98.3 (13.5) | 96.5 (15.1)
Statistical Analysis 1: Comparison: Exclusive Smokers vs Exclusive E-Cig Users vs Never Users; Test type: Other; p = .022, ANCOVA; Age, sex, and race/ethnicity were covaried. Test for group difference: F (2, 381) = 3.877, p = .022; Group difference tested after correction for false discovery rate at .05, therefore we followed with post-hoc pairwise comparisons
Statistical Analysis 2: Comparison: Exclusive E-Cig Users vs Never Users; Never Users minus Exclusive E-Cig Users; Test type: Other; p = 0.952, ANCOVA post-hoc pairwise group compariso; Age, sex, and race were covaried
Statistical Analysis 3: Comparison: Exclusive Smokers vs Never Users; post hoc pairwise group comparisons.. Never Users minus Exclusive Smokers; Test type: Other; p = 0.014, ANCOVA post-hoc pairwise group compariso; Age, sex, and race were covaried
Statistical Analysis 4: Comparison: Exclusive Smokers vs Exclusive E-Cig Users; Exclusive E-Cig Users minus Exclusive Smokers; Test type: Other; p = 0.011, ANCOVA post-hoc pairwise group compariso — Age, sex, and race were covaried

21. Secondary Outcome: Fractional Exhaled Nitric Oxide (FeNO)
Description: Fractional Exhaled Nitric Oxide is a measure of airway inflammation measured before an acute exposure challenge.
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Number analyzed (Participants) | 111 | 163 | 114
ppb | 9.7 (12.3) | 14.5 (14.7) | 16.2 (11)
Statistical Analysis 1: Comparison: Exclusive Smokers vs Exclusive E-Cig Users vs Never Users; Test type: Other; p < .001, ANCOVA; Age, sex, and race/ethnicity were covaried. Outcome variable log-transformed for analysis. Test for group difference: F (2, 381) = 33.442, p < .001; Group difference tested for false discovery rate at .05 and followed with post-hoc pairwise comparisons
Statistical Analysis 2: Comparison: Exclusive E-Cig Users vs Never Users; Never Users minus Exclusive E-Cig Users:; Test type: Other; p = 0.013, ANCOVA post-hoc pairwise group compariso; Age, sex, and race were covaried; Mean Difference (Final Values) = 0.180, 95% CI 2-sided [0.039 to 0.322] — Estimated marginal mean differences (log-transformed scale)
Statistical Analysis 3: Comparison: Exclusive Smokers vs Never Users; Never Users minus Exclusive Smokers; Test type: Other; p < 0.001, ANCOVA post-hoc pairwise group compariso; Age, sex and race were covaried; Mean Difference (Final Values) = 0.679, 95% CI 2-sided [0.514 to 0.844] — Estimated marginal mean differences (log-transformed scale)
Statistical Analysis 4: Comparison: Exclusive Smokers vs Exclusive E-Cig Users; Exclusive E-Cig users minus Exclusive Smokers; Test type: Other; p < 0.001, ANCOVA post-hoc pairwise group compariso; Age, sex, and race/ethnicity were covaried; Mean Difference (Final Values) = 0.498, 95% CI 2-sided [0.336 to 0.660] — Estimated marginal mean differences (log-transformed scale)"

22. Secondary Outcome: Autonomic Measures - RMSSD
Description: Root mean square of standard deviation of rr intervals. Obtained fasting and refraining from nicotine exposure using the Sphymocor system. We used 10 or more minutes of supine data to derive heart rate variability measures.
Time Frame: v2 was generally 1-2 weeks after enrollment visit, with a window up to 4 weeks from V1
Measure: Median (Inter-Quartile Range); unit: ms
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Number analyzed (Participants) | 105 | 158 | 105
ms | 43.6 [25.95 to 56.20] | 63.3 [40.60 to 89.50] | 58.3 [41.40 to 82.80]
Statistical Analysis 1: Comparison: Exclusive Smokers vs Exclusive E-Cig Users vs Never Users; Test type: Other; p = .150, ANCOVA; Age, sex, and race/ethnicity were covaried. Test for group difference: F (2, 361) = 1.904, p = .150

23. Secondary Outcome: Arterial Pulse Wave Analysis (PWA), Augmentation Index (at 75 Bpm, %)
Description: Analysis of radial pressure wave forms allows for non-invasive estimation of central aortic pressures, accounting for pressure amplification and the amplitude of the arterial pulse wave as it moves through arteries away from the heart. The Atcor Sphygmacor system can derive central aortic pressures from radial tracings using a validated transfer function. This computation is performed using the pulse wave analysis (PWA) mode. Pulse Wave Analysis via radial tonometry was obtained as a measure of chronic exposure.
Time Frame: v2 was generally 1-2 weeks after enrollment visit, with a window up to 4 weeks from V1
Measure: Median (Inter-Quartile Range); unit: percentage of central pulse pressure
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Number analyzed (Participants) | 117 | 161 | 114
percentage of central pulse pressure | 19.5 [7.25 to 29.00] | 0.50 [-8.50 to 12.00] | 1.00 [-9.00 to 11.13]
Statistical Analysis 1: Comparison: Exclusive Smokers vs Exclusive E-Cig Users vs Never Users; Test type: Other; p < .001, ANCOVA; Age, sex, and race/ethnicity were covaried. Test for group difference: F (2, 385) = 17.872, p < .001; Group difference tested for false discovery rate at .05, and followed with post-hoc pairwise comparisons. Estimated marginal mean differences:
Statistical Analysis 2: Comparison: Exclusive E-Cig Users vs Never Users; Never Users minus Exclusive E-Cig Users; Test type: Other; p = 0.003, ANCOVA post-hoc pairwise group compariso; Age, sex, and race were covaried; Mean Difference (Final Values) = -3.632, 95% CI 2-sided [-6.019 to -1.245]
Statistical Analysis 3: Comparison: Exclusive Smokers vs Never Users; Never Users minus Exclusive Smokers; Test type: Other; p < 0.001, ANCOVA post-hoc pairwise group compariso; Age, sex, and race were covaried; Mean Difference (Final Values) = -8.380, 95% CI 2-sided [-11.14 to -5.62]
Statistical Analysis 4: Comparison: Exclusive Smokers vs Exclusive E-Cig Users; Exclusive E-Cig Users minus Exclusive Smokers; Test type: Other; p = 0.001, ANCOVA post-hoc pairwise group compariso; Age, sex, and race were covaried; Mean Difference (Final Values) = -4.748, 95% CI 2-sided [-7.456 to -2.040]

24. Secondary Outcome: Exercise Treadmill Stress Test (ETT)-Peak METS
Description: An ETT to determine exercise capacity will be completed as a measure of chronic exposure. Peak metabolic equivalents (METs, 1 MET=3.5 ml O2 uptake/kg body weight/minute) were determined at all exercise stages, peak exercise, and 1-minute post-exercise.
Time Frame: Treadmill test done only once at the end of v2 after completion of all other post-challenge assessment tests. V2 was scheduled 1-4 weeks from enrollment vist
Measure: Mean (Standard Deviation); unit: METS
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Number analyzed (Participants) | 83 | 157 | 110
METS | 8.39 (3.19) | 10.29 (2.01) | 11.06 (2.42)
Statistical Analysis 1: Comparison: Exclusive Smokers vs Exclusive E-Cig Users vs Never Users; Test type: Other; p < .001, ANCOVA; Age, sex, and race/ethnicity were covaried. Test for group difference: F (2, 343) = 17.056, p < .001; Group difference tested for false discovery rate at .05, and followed with post-hoc pairwise comparisons
Statistical Analysis 2: Comparison: Exclusive E-Cig Users vs Never Users; Never Users minus Exclusive E-Cig Users; Test type: Other; p < 0.001, ANCOVA post-hoc pairwise group compariso; age, sex and race were covaried; Mean Difference (Final Values) = 1.279, 95% CI 2-sided [0.733 to 1.824]
Statistical Analysis 3: Comparison: Exclusive Smokers vs Never Users; Never Users minus Exclusive Smokers; Test type: Other; p < 0.001, ANCOVA post-hoc pairwise group compariso; Age, sex and race were covaried; Mean Difference (Final Values) = 1.739, 95% CI 2-sided [1.083 to 2.395]
Statistical Analysis 4: Comparison: Exclusive Smokers vs Exclusive E-Cig Users; Exclusive E-Cig Users minus Exclusive Smokers; Test type: Other; p = 0.165, ANCOVA post-hoc pairwise group compariso; age, sex and race were covaried; Mean Difference (Final Values) = 0.460, 95% CI 2-sided [-0.190 to 1.110]

25. Secondary Outcome: Diastolic Blood Pressure (DBP)
Description: During V2, Diastolic Blood Pressure was measured using the oscillometric technique before an acute exposure challenge following a standardized protocol. After resting supine for 10 minutes blood pressure was measured on both arms and the average of the last two values was used. Participants attended v2 in the morning, fasting and refraining from nicotine products for at least 8 hours.
Time Frame: V2 was generally 1-2 weeks after enrollment with a window up to 4 weeks from V1, recorded after resting supine for 10 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Number analyzed (Participants) | 115 | 164 | 114
mmHg | 76.6 (10.7) | 71.1 (7.5) | 70.4 (7.1)
Statistical Analysis 1: Comparison: Exclusive Smokers vs Exclusive E-Cig Users vs Never Users; Test type: Other; p = .199, ANCOVA; Age, sex, and race/ethnicity were covaried. Test for group difference: F (2, 386) = 1.621, p = .199

26. Secondary Outcome: Peak Rate Pressure Product (RPP, Peak Heart Rate Multiplied by Peak Systolic Blood Pressure)
Description: Peak RPP was calculated by multiplying maximun heart rate during exercise by systolic blood pressure as a reliable assessment of cardiac workload
Time Frame: During V2 (1-4 weeks after enrollment visit) the treadmill stress test was done last, following Nicotine-containing product challenge (users) or pretend 10 minute exposure for controls
Measure: Mean (Standard Deviation); unit: mmHg x bpm
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Number analyzed (Participants) | 84 | 157 | 110
mmHg x bpm | 249.99 (62.82) | 284.76 (51.36) | 290.86 (48.61)
Statistical Analysis 1: Comparison: Exclusive Smokers vs Exclusive E-Cig Users vs Never Users; Test type: Other; p < 0.001, ANCOVA; Age, sex, and race/ethnicity were covaried. Test for group difference: F (2, 343) = 17.056, p< .001; Group difference tested for false discovery rate at .05, and followed with post-hoc pairwise comparisons
Statistical Analysis 2: Comparison: Exclusive E-Cig Users vs Never Users; Never Users minus Exclusive E-Cig users; Test type: Other; p < 0.001, ANCOVA post-hoc pairwise group compariso; Age, sex and race were covaried; Mean Difference (Final Values) = 1.279, 95% CI 2-sided [0.733 to 1.824]
Statistical Analysis 3: Comparison: Exclusive Smokers vs Never Users; Never Users minus Exclusive Smokers; Test type: Other; p < 0.001, ANCOVA post-hoc pairwise group compariso; age, sex, race covaried; Mean Difference (Final Values) = 1.739, 95% CI 2-sided [1.083 to 2.395]
Statistical Analysis 4: Comparison: Exclusive Smokers vs Exclusive E-Cig Users; Exclusive E-Cig Users minus Exclusive Smokers; Test type: Other; p = 0.165, ANCOVA post-hoc pairwise group compariso; Age, sex and race were covaried; Mean Difference (Final Values) = 0.460, 95% CI 2-sided [-0.190 to 1.110]

27. Secondary Outcome: Heart Rate Reserve (%)
Description: Measure of maximal exercise capacity adjusted for age, calculated as max heart rate during treadmill divided by (220 minus the participant's age in yrs)
Time Frame: During V2 (1-4 weeks after enrollment visit) the treadmill stress test was done last, following Nicotine-containing product challenge (users) or 10 minute pretend exposure for never-users
Measure: Mean (Standard Deviation); unit: percentage of heart rate reserve
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Number analyzed (Participants) | 84 | 157 | 110
percentage of heart rate reserve | 83.25 (11.58) | 87.89 (8.81) | 91.72 (7.58)
Statistical Analysis 1: Comparison: Exclusive Smokers vs Exclusive E-Cig Users vs Never Users; Test type: Other; p < 0.001, ANCOVA; Age, sex, and race/ethnicity were covaried. Test for group difference: F (2, 343) = 17.056, p< .001; Group difference tested for false discovery rate at .05, and followed with post-hoc pairwise comparisons
Statistical Analysis 2: Comparison: Exclusive E-Cig Users vs Never Users; Never Users minus Exclusive E-Cig Users; Test type: Other; p < 0.001, ANCOVA post-hoc pairwise group compariso; Age, sex, race were covaried; Mean Difference (Final Values) = 1.279, 95% CI 2-sided [0.733 to 1.824]
Statistical Analysis 3: Comparison: Exclusive Smokers vs Never Users; Never Users minus Exclusive Smokers; Test type: Other; p < 0.001, ANCOVA post-hoc pairwise group compariso; Age, sex and race were covaried; Mean Difference (Final Values) = 1.739, 95% CI 2-sided [1.083 to 2.395]
Statistical Analysis 4: Comparison: Exclusive Smokers vs Exclusive E-Cig Users; Exclusive E-Cig Users minus Exclusive Smokers; Test type: Other; p = 0.165, ANCOVA post-hoc pairwise group compariso; Age, sex and race were covaried; Mean Difference (Final Values) = 0.460, 95% CI 2-sided [-0.190 to 1.110]

28. Secondary Outcome: 60 Seconds Heart Rate Recovery (Beats Per Minute)
Description: Difference in heart rate 60 seconds post treadmill minus maximal heart rate during treadmill..
Time Frame: as for outcome 26
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
Number analyzed (Participants) | 84 | 157 | 110
beats per minute (bpm) | 19.62 (10.38) | 26.74 (9.06) | 28.06 (8.26)
Statistical Analysis 1: Comparison: Exclusive Smokers vs Exclusive E-Cig Users vs Never Users; Test type: Other; p < 0.001, ANCOVA; Age, sex, and race/ethnicity were covaried. Test for group difference: F (2, 344) = 10.075, p < .001; [other analysis details as in outcome 23, analysis 1]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Exclusive Smokers | Exclusive E-Cig Users | Never Users
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/164 | 0/114
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/164 | 0/114
Other Adverse Events (participants affected / at risk) | 0/117 | 1/164 | 1/114
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exclusive Smokers (N=117) | Exclusive E-Cig Users (N=164) | Never Users (N=114)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — one e-cigarette user felt transient nausea after vaping
Vasovagal response (General disorders) | 0 (0) | 0 (0) | 1 (1) — During blood draw a control subject fainted. Recovered in a few seconds but then vomited. Remained in observation for 30 minutes afterwards until all symptoms subsided

LIMITATIONS AND CAVEATS:
Observational study, changes observed with product challenge are not proof of the causal effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT03863509/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT03863509/ICF_001.pdf